CLINICAL TRIAL: NCT03731845
Title: Evaluation of Individual Sensitivity to the Gonadotoxicity of Chemotherapy in Young Patients With Breast Cancer
Acronym: ESIGON
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: K160913J; 2017-A02111-52 (Other: ID-RCB)
Record Dates: First submitted 2018-08-10; First posted 2018-11-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; ovarian reserve; primary ovarian insufficiency; chemotherapy; single nucleotide polymorphism
MeSH Terms: conditions — Breast Neoplasms; Primary Ovarian Insufficiency | interventions — Blood Specimen Collection; Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient (Experimental)
  Interventions: Genetic: Blood sample for genetic test; Biological: Blood sample for hormonal measurement; Other: Ovarian ultrasound scan

INTERVENTIONS:
Genetic: Blood sample for genetic test — Patients will be genotyped for single nucleotide polymorphism previously found to be associated with age at natural menopause
Biological: Blood sample for hormonal measurement — at each visit : 2x7ml. At the end of the study hormonal measurements (AMH, P4, LH, FSH, E25)
Other: Ovarian ultrasound scan — Ovarian ultrasound scan at follow up visits (Y1,Y1.5, Y2.5 Y3.5 Y4.5 Y5.5)

SUMMARY:
Over the past decade, advances in diagnosis and treatments have dramatically increased the rates of cure for young patients with cancer. As a consequence, a new population of cancer survivors has emerged whose fertility is compromised after cancer therapy. Indeed, gonadotoxicity is a well-known long-term side effect of cancer treatment in young patients having survived malignant diseases. More than 80% of women of childbearing age, treated for breast cancer with standard protocol of neoadjuvant (4 cycles of 5-fluorouracile - epirubicin- cyclophosphamide (FEC) and 4 cycles of docetaxel) or adjuvant chemotherapy (3 FEC and 3 docetaxel), show an alteration of their ovarian reserve 2 years after completion of the treatment, as a result of chemotherapy-related follicular loss. Therefore, according to the extent of the follicular damages, the gonadal function may vary from moderate to severe diminished ovarian reserve (DOR) and possibly to the ultimate stage of premature ovarian insufficiency (POI).

Investigators propose a multicentric and prospective study of a cohort of young women with breast cancer to evaluate whether genetic polymorphisms, previously identified as being correlated with age at menopause in the healthy population, are associated with the intensity of the follicular decline following chemotherapy in young breast cancer survivors.

DETAILED DESCRIPTION:
With 48 763 new cases in 2012, breast cancer represents the first female cancer in France. Although the incidence of this malignancy peaks after the age of 60 years, nearly 2500 of reproductive-age women are diagnosed with breast cancer every year. Recent advances in cancer therapy markedly improved the rates of cure for young adult suffering from cancers. Over the past decade, the mortality rates in breast cancer patients has decreased by more than 1.6% per year. The five year survival rate for women under 45 with breast cancer is now approaching 80%. As a consequence, a new population of young cancer survivors has emerged whose fertility is compromised after cancer therapy. Thus, the question of fertility preservation (FP) in young cancer patients has become a major issue in the care-personalized path. Indeed, information regarding the risks of infertility and FP counselling may contribute to improving the quality of life and the coping of patients with the burden of cancer treatment. Therefore, oncofertility counselling by a specialist is now recommended for all young cancer patients having to undergo treatment that may reduce the fertility potential.

Gonadotoxicity is a well-known long-term side effect of cancer treatment in young patient having survived malignant diseases. Neoadjuvant or adjuvant chemotherapy usually combining alkylating agent and taxane, is often recommended for young women presenting with breast cancer. However, alkylating agents, such as cyclophosphamide have been shown to cause extensive dose-dependent loss of primordial follicles in cancer patients. Beside a enhancement of apoptosis, cyclophosphamide might induce a follicular loss through an activation of the primordial follicle recruitment: the "burnout" phenomenon.

Moreover, the extent of ovarian damages depends not only on the nature and dose of chemotherapy but also on age and ovarian reserve before treatment. Women age at chemotherapy administration is one of the most predictive risk factor of follicular depletion after the end of treatment. Therefore, according to the extent of the follicular damages, the gonadal function may vary from moderate to severe diminished ovarian reserve (DOR) and possibly to the ultimate stage of premature ovarian insufficiency (POI).

Currently, patients' age and the values of markers of the follicular ovarian status (serum anti-Müllerian hormone (AMH) levels and ultrasonographic antral follicle count (AFC), measured before the initiation of gonadotoxic treatment, are considered the most accurate predictive factors of post chemotherapy ovarian function. However, they may have some limitations since important inter-individual variations in the ovarian reserve two years after completion of treatment are reported in patients displaying similar age, AMH as well as AFC. This observation suggests that, besides environmental and pathologic variables, genetic variations, inducing different ovarian sensitivity to chemotherapy, might be at play.

Indeed, in healthy women, age at natural menopause varies from 40 to 55 years and is characterized by a strong familial concordance. Many studies of large genome-wide association (GWAS) found a link between the age and variants of some genes involved in DNA repair, DNA maintenance and folliculogenesis as initial follicular recruitment. Since these genes may have an influence on the ovarian reserve (together with the effects of gonadotoxic treatment regimens), investigators hypothesize that genetic polymorphisms known to be associated with age at menopause (BRSK1 (rs1 172822), ARHGEF7 (rs7333181), MCM8 (rs236114), PCSK1 (rs271924), IGF2R (rs9457827), TNF (rs909253), AMH (rs10407022) and AMHR2 (rs2002555) could be linked to the intensity of the follicular depletion after chemotherapy.

The primary objective is to evaluate whether genetic polymorphisms, previously identified as being correlated with age at menopause onset in the healthy population, are associated with the intensity of the follicular decline following chemotherapy in young breast cancer survivors.

The secondary objectives are to evaluate the association between genetic polymorphisms and other parameters related to female fertility, as menstrual cycle profile, pregnancy rate, serum anti-mullerian hormone (AMH) levels and ultrasonographic antral count (AFC) after chemotherapy such as the menstrual cycle profile and pregnancy rates.

Eligible subjects followed in the different participating centers will be included in this study. Informed consent will be obtained from all participating individuals before blood sample collection and molecular studies. AMH measurement and AFC will be performed before the cancer treatment randomly during the menstrual cycle phase. In the same time, blood samples will be taken for the genotyping. All patients will receive adjuvant or neoadjuvant chemotherapy containing cyclophosphamide, epirubicin, 5-FU and docetaxel. Patients will be evaluated 12 and 24 months after the end of the treatment. A clinical (menstrual cyclicity) and hormonal (AMH, FSH) evaluation associated with ultrasound evaluation of AFC of enrolled patients will be performed. Thus, association between genetic polymorphism and the depth of ovarian decline (classified as: normal ovarian reserve, moderate DOR, severe DOR or POI) after healing will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 36 years
* Diagnosis of breast cancer
* BMI≤30 Kg/m2
* Baseline antral Follicular count (before initiation of chemotherapy): 10-40 follicles measuring 2 - 9 mm in diameter
* Regular and ovulatory menstrual cycles
* Indication of neoadjuvant (4 FEC and 4 docetaxel) or adjuvant (3 FEC and 3 docetaxel) chemotherapy
* Free informed and written consent, dated and signed by the patient and the investigator
* Patient affiliated to the French National Social Security System

Non inclusion criteria

* Previous history of chemotherapy
* History of ovarian surgery or endometrioma
* Ovarian Polycystic Syndrome
* DOR or POI before chemotherapy
* Virgin patients

Exclusion Criteria:

- Intensification of chemotherapy

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 73 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of ovarian reserve | 5 years after completion of chemotherapy
  is an aggregated measure of FSH, AMH serum level, Antral Follicle Count and menstrual profile :
  * Normal ovarian reserve: persistence of menstrual cycle, FSH<40 IU/L and AMH>1.1 ng/mL or AFC>7 follicles
  * Moderate diminished ovarian reserve : persistence of menstrual cycle, FSH<40 IU/L and 0.5≤AMH≤1.1 ng/mL or 5≤AFC≤7 follicles
  * Severe diminished ovarian reserve : persistence of menstrual cycle and AMH<0.5 ng/mL or AFC<5 follicles
  * Premature ovarian insufficiency is defined by amenorrhea above four months and FSH level ≥40 IU/L in women before 40 years.
  AMH serum levels and ultrasonographic evaluation of AFC will be evaluated FIVEyears after the end of chemotherapy.

SECONDARY OUTCOMES:
Menstrual profile: amenorrhea, spaniomenorrhea, normal cycle length (28-35 days) | 5 years
  To evaluate the association between genetic polymorphisms and other parameters related to female fertility after chemotherapy such as the menstrual cycle profile. These data will be obtained from clinical interrogatory performed by medical doctors.
Pregnancy rates | 5 years
  These data will be obtained from clinical interrogatory performed by medical doctors.
AMH level | 6, 12, 24, 36, 48, 60 months following the end of chemotherapy.
  To assess the evolution of ovarian reserve tests at the end of chemotherapy AMH level will be performed before the initiation of chemotherapy and 6, 12, 24, 36, 48, 60 months following the end of chemotherapy.
Antral Follicle Count (Ultrasound evaluation) | 6, 12, 24, 36, 48, 60 months following the end of chemotherapy.
  To assess the evolution of ovarian reserve tests at the end of chemotherapy Measurements of ultrasonographic AFC will be performed before the initiation of chemotherapy and 6, 12, 24, 36, 48, 60 months following the end of chemotherapy.
Follicular decline (definition below) | 2 years after the completion of chemotherapy
  A follicular decline will be defined as a moderate/severe DOR or a POI

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte SONIGO, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Michael Grynberg, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Antoine Béclère Hospital, Clamart, France

IPD SHARING:
Plan to Share IPD: Undecided